CLINICAL TRIAL: NCT06497036
Title: Multicenter Randomized Controlled Study of Efficacy, Safety and Immunogenicity of GP40141 (GEROPHARM, Russia) Compared With Nplate® (Amgen, the Netherlands) in Patients With Persistent or Early Immune Thrombocytopenia
Brief Title: Study of Efficacy, Safety and Immunogenicity of GP40141 (GEROPHARM, Russia) in Patients With Immune Thrombocytopenia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Geropharm (Industry)
Collaborators: Pharm-Holding (Unknown); I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GP40141-P4-03-02
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2023-10

CONDITIONS: Drug Effect; Safety Issues; Immunogenicity
Keywords: romiplostim, nplate, bioequivalence
MeSH Terms: interventions — romiplostim

STUDY DESIGN:
Intervention Model Description: Multicenter, single-blind, randomized controlled trial of efficacy and safety in two parallel groups
Who Masked: Participant
Masking Description: patients will not have access to the treatment assignment code and, therefore, will not know which study drug they are receiving
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP40141 (Experimental): Lyophilized powder for solution 250 mcg in vials is diluted in sterile water for injection to a concentration of 500 mcg/ml. Administer once a week.
  Cohort 1 Starting dose of romiplostim is 1 mcg/kg actual body weight. The weekly dose of romiplostim is increased in increments of 1 mcg/kg body weight until the patient's platelet count reaches ≥50 x 10*9/L. Platelet counts are assessed weekly.
  Cohort 2
  * For subjects receiving Nplate®, a switch to GP40141 at an equivalent dose is recommended 7±2 days after the last Nplate® administration. The transition is equidosal since the drugs contain the same active ingredient.
  * For patients receiving eltrombopag or Etrombopag-29F® (Pharmproekt, Russia)), it is recommended to switch to GP40141 at an initial dose of 1 mcg/kg the day after the last dose of eltrombopag.
  The maintenance dose, dose adjustment, and maximum dose are consistent for both cohorts. Duration of therapy with study drugs will be 26 weeks.
  Interventions: Drug: GP404141
- Nplate (Active Comparator): Lyophilized powder for solution 250 mcg in vials is diluted in sterile water for injection to a concentration of 500 mcg/ml. Administer once a week.
  Cohort 1 Starting dose of romiplostim is 1 mcg/kg actual body weight. The weekly dose of romiplostim is increased in increments of 1 mcg/kg body weight until the patient's platelet count reaches ≥50 x 10*9/L. Platelet counts are assessed weekly.
  Cohort 2
  Initial dose:
  • For patients receiving eltrombopag or Etrombopag-29F® (Pharmproekt, Russia)), it is recommended to switch to at Nplate® initial dose of 1 mcg/kg the day after the last dose of eltrombopag.
  The maintenance dose, dose adjustment, and maximum dose are consistent for both cohorts. Duration of therapy with study drugs will be 26 weeks.
  Interventions: Drug: Nplate

INTERVENTIONS:
Drug: GP404141 — subcutaneous injection
  Other Names: romiplostim
  Arms: GP40141
Drug: Nplate — subcutaneous injection
  Other Names: romilostim
  Arms: Nplate

SUMMARY:
The goal of this clinical trial is to demonstrate equivalent efficacy and comparable safety of the drug GP40141 (GEROPHARM, Russia) in comparison with the drug Nplate® (Amgen, the Netherlands). the main questions are

1. Assess the effectiveness of GP40141 in comparison with Nplate®.
2. Assess the immunogenicity of GP40141 in comparison with the drug Nplate®.
3. Assess the safety of GP40141 in comparison with the drug Nplate®.
4. Assess the safety of changing romiplostim and eltrombopag to GP40141.
5. Assess the pharmacokinetic parameters of the study drugs in patients with primary immune thrombocytopenia.

Participants divided into 2 cohorts (naïve or treated with a thrombopoietin receptor agonist) will receive romiplostim and platelet response, immune response and adverse reactions will be assessed.

DETAILED DESCRIPTION:
The study will be conducted in adult patients with persistent or chronic primary immune thrombocytopenia. Patients both naïve to treatment with a thrombopoietin receptor agonist (cohort 1) and those who have previously received therapy (cohort 2) will be included.

Cohort 1:

Adult steroid-dependent or steroid-refractory patients with persistent or chronic primary immune thrombocytopenia (PIT) with or without a history of splenectomy who have not previously received thrombopoietin receptor agonist (TPO-RA) therapy.

Cohort 2:

Adult patients with persistent or chronic primary immune thrombocytopenia receiving TPO-RA (romiplostim or eltrombopag) for ≥12 weeks and with sustained response status at screening.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.
* male or female
* Age ≥18 years
* Diagnosis of primary immune thrombocytopenia (PIT).
* Duration of PIT at the Screening Visit: for cohort 1: ≥3 months; for cohort 2: ≥6 months.
* PIT therapy with glucocorticosteroids (GCS) for cohort 1: duration of continuous therapy ≥3 months at the Screening Visit or ≥2 courses of pulse therapy during the year before the Screening Visit;
* TPO-RA therapy: for cohort 1: no history of TPO-RA use; for Cohort 2: Use of TPO-RA for ≥12 weeks at the Screening Visit;
* No increase in TPO-RA dose during the 4 weeks preceding the end of screening.
* Blood platelet count: for cohort 1: mean platelet count ≤30×10*9/L, based on the last two measurements 7±2 days apart, each of which had a platelet count ≤35×10*9/L OR steroid dependence, defined as the use of prednisolone at a daily dose of >5 mg (or another corticosteroid at an equivalent dose) for ≥2 months before the Screening Visit to maintain a platelet count ≥30×10*9/L OR to prevent bleeding; for cohort 2: platelet count ≥50×10*9/ml for ≥6 weeks out of the last 8 weeks of follow-up with platelet counts every 7±2 days and no emergency treatment for severe hemorrhagic syndrome in the last 12 weeks before the Screening Visit.
* Consent and ability to comply with the procedures of the Protocol, as well as the prohibitions and restrictions provided for by the Research Protocol.

Exclusion Criteria:

* Hypersensitivity to romiplostim.
* History of TPO-RA use: for cohort 1: any TPO-RA; for cohort 2: any TPO-RA, with the exception of romiplostim and eltrombopag.
* Unpromising treatment with romiplostim in the opinion of the Researcher
* Splenectomy <24 weeks prior to the Screening Visit or planned splenectomy during the study.
* Treatment with rituximab within the 14 weeks preceding the Screening Visit, or planned treatment with rituximab during the study.
* Treatment with intravenous immunoglobulin or anti-D immunoglobulin during the 2 weeks preceding the Screening Visit, or planned use during the study.
* Therapy with hematopoietic growth factors during the 4 weeks preceding the Screening Visit, or their planned use during the study.
* Therapy with alkylating chemotherapy drugs during the 8 weeks preceding the Screening Visit, or their planned use during the study.
* Use of other medicines listed in section 5.3.3. of this study protocol.
* Participation in a clinical trial of an investigational drug or investigational medical device within 4 weeks or 5 half-lives (whichever is longer) preceding the Screening Visit.
* Secondary immune thrombocytopenia in the following diseases: autoimmune thyroiditis, systemic lupus erythematosus (SLE), antiphospholipid syndrome (APLS), lymphoproliferative diseases, drug-mediated, viral origin (herpes viruses, HIV, chronic viral hepatitis).
* Hereditary thrombocytopenia.
* Diseases of the hematopoietic system accompanied by thrombocytopenia (for example, acute leukemia, aplastic anemia, myelodysplastic syndrome, lymphoproliferative diseases).
* Metastatic bone marrow lesions.
* Uncontrolled concomitant diseases of internal organs.
* Arterial thrombosis (for example, myocardial infarction, acute cerebrovascular accident) within 1 year preceding the Screening Visit.
* History of venous thrombosis.
* High risk of venous thrombosis and thromboembolism, defined as the presence of at least three of the following risk factors:
* diabetes;
* smoking;
* use of combined oral contraceptives or menopausal hormone therapy;
* positive titer of antiphospholipid antibodies;
* hypercholesterolemia (>240 mg/dl or >13 mmol/l);
* hypertriglyceridemia;
* arterial hypertension requiring therapy.
* HIV infection.
* Viral hepatitis B or C.
* Oncological and/or oncohematological disease beyond the stage of complete 5-year remission at the Screening Visit.
* Major surgery ("major surgery") within 8 weeks preceding the Screening Visit, or incomplete recovery from surgery at the Screening Visit.
* Pregnancy or lactation in women.
* Hospitalization for any reason planned during the patient's participation in the study.
* A history of mental disorders that do not allow you to adequately assess your behavior and follow the conditions of the study protocol.
* Alcoholism. Alcoholism or consumption of alcohol in quantities exceeding for men: 14 units. per week (on average); for women: 7 units. per week (on average).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with platelet response | 10 weeks
  Blood platelet count ≥50×10*9/L after 10 weeks of therapy (at Visit 11), or blood platelet count ≥200×10*9/L at the last assessment if the study was terminated early.
Number of adverse events (AEs) | 10 weeks
  AEs including ones of special interest: bleeding, thrombotic and thromboembolic events.
Proportion of subjects experiencing AEs, | 10 weeks
  AEs including ones of special interest: bleeding, thrombotic and thromboembolic events.
Proportion subjects with a immune response to romiplostim | 26 weeks
  Proportion of initially immunonaive subjects with a documented immune response to romiplostim at Visits 8 and 26 (weeks 8 and 26).
Proportion subjects with a immune response to endogenous thrombopoietin | 26 weeks
  Proportion of initially immunonaive subjects with a documented immune response to endogenous thrombopoietin at Visits 8 and 26 (weeks 8 and 26).

CONTACTS AND LOCATIONS:
Overall Officials: Bulat Bakirov, MD, Principal Investigator — Bashkir State Medical University of the Ministry of Health of the Russian Federation; Elena Borisenkova, Principal Investigator — Kaluga Regional Clinical Hospital; Olga Vinogradova, Principal Investigator — City Clinical Hospital named after S.P. Botkin of the Moscow City Health Department; Igor Davydkin, Principal Investigator — Samara State Medical University of the Ministry of Health of the Russian Federation; Dmitry Kirtbaya, Principal Investigator — Oncological dispensary No. 2 of the Ministry of Health of the Krasnodar Territory; Galina Salogub, Principal Investigator — National Medical Research Center VA Almazov Ministry of Health of the Russian Federation
Locations (6):
- Russia (6):
  - Kaluga Regional Clinical Hospital, Kaluga
  - City Clinical Hospital S.P. Botkin of the Moscow City Health Department, Moscow
  - National Medical Research Center in name of V.A. Almazov " of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Samara State Medical University" of the Ministry of Health of the Russian Federation, Samara
  - Oncological dispensary No. 2 of the Ministry of Health of the Krasnodar Territory, Sochi
  - Federal State Budgetary Educational Institution Bashkir State Medical University of the Ministry of Health of the Russian Federation, Ufa

REFERENCES:
- [Derived] Melikyan AL, Protsenko EA, Salogub GN, Bakirov BA, Davydkin IL, Kovalik VV, Gefen ML, Matvienko YD, Saparova VB, Khokhlov AL, Makarenko IE, Drai RV. Multicenter Single-Blind Randomized Controlled Trial of the Romiplostim Biosimilar. EJHaem. 2025 Jul 24;6(4):e70105. doi: 10.1002/jha2.70105. eCollection 2025 Aug. PMID 40708707